CLINICAL TRIAL: NCT00610350
Title: Levosimendan Pre-Treatment in Patients Undergoing Coronary Artery Bypass Graft Surgery: a Double-Blind, Single Center, Prospective, Randomized, Placebo-Controlled Trial
Brief Title: Levosimendan and Myocardial Protection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University College London Hospitals (Other)
Responsible Party: Vincenzo De Santis, University of Rome "Sapienza"
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LV 2003; LV-2003-01
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-01

CONDITIONS: Myocardial Protection
Keywords: Levosimendan; pre-conditioning; cardiac surgery; myocardial function; contractility; heart; ischaemia
MeSH Terms: conditions — Ischemia | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L (Experimental)
  Interventions: Drug: levosimendan
- P (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levosimendan — 24 μg/kg administered as a slow i.v. 50 ml bolus through the central venous port of a pulmonary artery catheter over the 10 minutes before initiation of CPB
  Arms: L
Drug: Placebo — an identical-appearing placebo prepared and labelled by the pharmacy was administered as a slow i.v. 50 ml bolus through the central venous port of a pulmonary artery catheter over the 10 minutes before initiation of CPB
  Arms: P

SUMMARY:
The aim of this study is to investigate whether pharmacological pre-treatment with levosimendan reduces intensive care unit (ICU) length of stay in patients undergoing elective myocardial revascularization under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* intention to perform first-time multi-vessel CABG

Exclusion Criteria:

* unstable angina
* valvular disease
* diabetes mellitus treated with sulphonylurea drugs
* renal failure
* severe hepatic disease
* severe chronic obstructive pulmonary disease
* a history of prior CABG surgery
* recent myocardial infarction (MI) within the previous month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Length of ICU stay | two weeks

SECONDARY OUTCOMES:
Length of hospital stay | 3 weeks
Tracheal intubation time | one week
Inotropic support over the first 7 days | one week

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo De Santis, M.D., Principal Investigator — University of Roma La Sapienza
Locations (1):
- University of Rome "Sapienza", Rome, Italy

REFERENCES:
- [Derived] Tritapepe L, De Santis V, Vitale D, Guarracino F, Pellegrini F, Pietropaoli P, Singer M. Levosimendan pre-treatment improves outcomes in patients undergoing coronary artery bypass graft surgery. Br J Anaesth. 2009 Feb;102(2):198-204. doi: 10.1093/bja/aen367. PMID 19151048